CLINICAL TRIAL: NCT03892785
Title: MEthotrexate Versus TOcilizumab for Treatment of GIant Cell Arteritis: a Multicenter, Randomized, Controlled Trial
Acronym: METOGiA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BONNOTTE PHRC N 2017
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab group (Experimental)
  Interventions: Drug: Prednisone treatment; Drug: Tocilizumab treatment; Other: Questionnaires; Biological: Blood samples
- Methotrexate group (Active Comparator)
  Interventions: Drug: Prednisone treatment; Drug: Methotrexate treatment; Other: Questionnaires; Biological: Blood samples

INTERVENTIONS:
Drug: Prednisone treatment — tapering prednisone regimen
Drug: Tocilizumab treatment — Tocilizumab 162 mg/week subcutaneous from W0 to W51 (52 injections)
  Arms: Tocilizumab group
Drug: Methotrexate treatment — Methotrexate subcutaneous from W0 to W51 (52 administrations).
  * W0: 7.5 mg/week
  * W1: 0.2 mg/Kg/week
  * W2 to W51: 0.3 mg/Kg/week (without exceeding 20 mg/week) Folic acid 10 mg/week, 48h after taking Methotrexate, from W0 to W51
  Arms: Methotrexate group
Other: Questionnaires — HAQ, SF-36, FACIT-fatigue
Biological: Blood samples — Additionnal blood samples for immunomonitoring

SUMMARY:
Giant-cell arteritis (GCA) is the most frequent vasculitis after 50 years. It is characterized by a granulomatous inflammation of the wall of large vessels, involving especially the aorta and extra-cranial branches of the external carotid, with vascular remodelling leading to ischemic manifestations such as temporal headaches, jaw claudication, scalp tenderness and visual loss. Most patients with GCA also present signs of systemic inflammation, including weight loss, fatigue and fever, together with an increased erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP) level.

Glucocorticoids (GC) are the cornerstone of the treatment of GCA. They are very effective and are usually given for 18-24 months to avoid relapses. Therefore, most patients develop GC-related complications that cause morbidity and disability. GC sparing strategies are thus required to improve the treatment of GCA.

* A 12-month treatment with tocilizumab (TCZ) has recently been shown to be effective in inducing and maintaining remission of GCA, with a dramatic GC-sparing effect. However, TCZ is an expensive drug; TCZ suppresses CRP synthesis and ESR elevation so that it is difficult to monitor patients; and importantly around 40% of patients relapse within 6 months after TCZ discontinuation, whether prescribed for 12 months or 4 months.
* In association with 6 months of prednisone, 10 mg/week of methotrexate (MTX) for 24 months lowers the risk of relapse at 24 months from 84% to 45%.

Therefore, the hypothesis is that 12 months of MTX treatment (0.3 mg/Kg/week, without exceeding 20 mg/week) is not inferior to 12 months of TCZ (162 mg SC/week) in term of prevention of relapse at 18 months. The MTX strategy might be more cost effective than TCZ.

In the present study, it is proposed to compare MTX versus TCZ in a multicenter randomized controlled trial. Moreover, the economic consequences associated with the use of MTX rather than TCZ will be also assess.

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Affiliation to a social security system
* Diagnosis of GCA, as defined by the revised GCA diagnosis criteria:44

  * Age ≥50 years at disease onset
  * AND History of erythrocyte sedimentation rate (ESR) ≥50 mm/h OR CRP≥20 mg/L (not mandatory if TAB is positive: see below)
  * AND At least one of the following:
* unequivocal cranial symptoms of GCA (new onset headache, scalp tenderness, jaw claudication, temporal artery abnormality, ischemia-related vision loss)
* unequivocal symptoms of polymyalgia rheumatica (PMR)

  o AND At least one of the following:
* Temporal artery biopsy (TAB) compatible with the diagnosis of GCA (non-necrotizing vasculitis with a predominance of mononuclear cell infiltration or granulomatous inflammation, usually with multinucleated giant cells)
* Evidence of large vessel vasculitis (aorta and/or epiaortic arteries):

  * angio-CT or angio-MRI: thickened arterial wall (≥2mm for the aorta and ≥1mm for epiaortic arteries) and/or contrast-enhanced arteries in T1-weighted sequences
  * PET scan: grade 3 tracer uptake of the arterial wall (grade 3 = arterial SUVmax superior to the SUVmax of the liver)
* Active GCA within 6 weeks before randomization. Active GCA is defined by ESR ≥30 mm/h or CRP ≥10 mg/L and at least one of the following:

  * ≥1 unequivocal cranial symptom(s) of GCA (new onset localized headache, scalp or temporal artery tenderness, ischemia-related vision loss, or otherwise unexplained mouth or jaw pain upon mastication)
  * ≥1 unequivocal symptom(s) of PMR, defined as shoulder and/or hip girdle pain associated with inflammatory stiffness
  * any other feature(s) judged by the clinical investigator to be consistent with GCA or PMR flares

Exclusion Criteria:

* Uncontrolled psychotic state
* Patient unable to give his/her consent
* Premenopausal women (menopause is defined as amenorrhea for more than 12 consecutive months)
* Non-compliant patients
* Weight<40 Kg or >100Kg
* Patients under maintenance of justice, wardship or legal guardianship
* History of intoxication (alcohol or medication) requiring hospitalization within 12 months before inclusion
* Current chronic alcohol abuse (consumption > 20g/day)
* Recent or incoming surgery within 12 months after inclusion
* History of stem cell or organ transplantation (except corneas performed more than 3 months prior inclusion)
* Primary or secondary immunodeficiency
* Hypersensitivity to methotrexate or tocilizumab, one of its excipients or another human or murine monoclonal antibody
* History of diverticulitis, inflammatory bowel disease, or other symptomatic gastrointestinal tract condition that might predispose to bowel perforation
* Patient refusing to sign methotrexate safety contract
* Prior treatment with any of the following:

  * Tocilizumab or methotrexate within 12 weeks before inclusion
  * Treatment with rituximab or other anti-CD20 agent within one year before inclusion
  * Treatment with cyclophosphamide within one year before inclusion
  * Hydroxychloroquine, cyclosporine A, dapsone, azathioprine, mycophenolate mofetil or janus kinase inhibitors within 4 weeks before inclusion
  * Tumor necrosis factor inhibitors within 8 weeks (infliximab) or 2 weeks (adalimumab or etanercept) before inclusion
  * Anakinra within 1 week before inclusion
* Long-term systemic glucocorticoid therapy ((except dermocorticoids and inhaled corticoids) for other conditions than GCA or PMR
* Patient with ≥3 prior glucocorticoid systematic therapies for another disease than GCA or PMR within the 6 months before inclusion
* Long-term treatment with sulfamethoxazole/trimethoprim (Bactrim®)
* Live vaccine administered within 30 days before inclusion
* Laboratory abnormalities:

  * AST or ALT >1.5 x upper limit of normal (ULN)
  * total bilirubin >ULN
  * platelets<100 G/L
  * leukocytes <3 G/L
  * neutropenia <1.5 G/L
  * lymphopenia <0.5 G/L
  * haemoglobin <8 g/dL (not related to GCA activity)
  * clearance of creatinine <30 ml/min/1,73 m2 [CKD EPI 2009]
  * positive HBs antigen or positive HCV antibodies
* Infections:

  * History of viral hepatitis B or C (chronic or acute)
  * HIV infection
  * Persistent infection or severe infection requiring hospitalization or intravenous antibiotics within 30 days before inclusion (antibiotic treatment tests are allowed, regardless of duration and route of administration)
  * Proven infection requiring oral antibiotics within 14 days before inclusion (antibiotic treatment tests are allowed, regardless of duration and route of administration)
  * Prior history of histoplasmosis or listeriosis
  * Active tuberculosis
  * Latent tuberculosis (diagnosis based on history of non-treated contact, opacity with a diameter greater than 1 cm on chest radiography, or positive in vitro test: Quantiferon Gold® or T-Spot-TB®).

NB: a history of tuberculosis for which treatment is over and was correctly precribed regarding usual recommendations is not an exclusion criteria, whatever the results of Quantiferon Gold® or T-Spot-TB® tests.

- Unstable or poorly controlled, acute or chronic disease, not due to GCA, and which contraindicates tocilizumab or methotrexate:

* Recurrent infections, unstable ischemic heart disease, renal failure (creatinine clearance <30 ml/min/1,73 m2 [CKD EPI 2009]), liver failure, current liver disease, heart failure ≥ NYHA stage III/IV, respiratory failure
* Neoplasia < 5 years, (except for in situ cervical cancer and skin carcinoma, except melanoma, with R0 resection)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients alive without relapse after initial remission or deviation from the scheduled regimen of prednisone | Week 78

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France

REFERENCES:
- [Derived] Lavergne A, Dumont A, Deshayes S, Boutemy J, Maigne G, Silva NM, Nguyen A, Gallou S, Philip R, Aouba A, de Boysson H. Efficacy and tolerance of methotrexate in a real-life monocentric cohort of patients with giant cell arteritis. Semin Arthritis Rheum. 2023 Jun;60:152192. doi: 10.1016/j.semarthrit.2023.152192. Epub 2023 Mar 20. PMID 36963127